CLINICAL TRIAL: NCT03482570
Title: Activity Behaviours in Patients With Malignant Pleural Effusion: Relationships With Quality of Life, and Respiratory Symptoms, and Survival
Brief Title: Activity Behaviours in Patients With Malignant Pleural Effusion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The University of Western Australia (Other); Edith Cowan University (Other); Queen Elizabeth Hospital, Hong Kong (Other); Princess Margaret Hospital, Hong Kong (Other Government); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. David Chi-leung Lam, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: HKU_UW_17_516
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Malignant Pleural Effusion
Keywords: Activity behaviors; Malignant pleural effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ActiGraph — Activity behaviours will be objectively assessed by 7-day triaxial accelerometer assessment (ActiGraph GT3X+ Pensacola, FL, USA). Participants will be asked to wear an accelerometer around their waist, 24 hours a day for 7 days.

SUMMARY:
The purpose of this research is to objectively assess activity behaviours (i.e., physical activity and sedentary behaviour) in patients with malignant pleural effusion. First, we aim to describe the physical activity and sedentary behavior of patients with MPE in Hong Kong. Secondarily, we aim to assess the relationships between activity behaviours and survival, quality of life, and respiratory symptoms e.g. shortness of breath.

DETAILED DESCRIPTION:
The development of a malignant pleural effusion (MPE) can be a consequence of metastatic spread of any cancer, but most commonly lung, breast and gynecological cancers or from primary pleural neoplasms (e.g., mesothelioma). The presence of MPE represents incurable disease and median survival ranges from 3 to 12 months from first presentation. Breathlessness is a common and debilitating symptom reported by this patient group and interventions are aimed at managing symptoms for optimal quality of life.

Breathlessness and other symptoms that result from MPE are likely to limit a person's ability to be physically active. Activity behaviours encompasses physical activity behaviour (i.e., low intensity physical activity and moderate-to-vigorous physical activity) and sedentary behaviour (i.e., sitting or reclining activities low in energy expenditure) accumulated during waking hours. Performance status measures are routinely used in cancer populations and are largely based on self-reported activity behaviors. While performance status is a reliable predictor of survival in patients with MPE, such measures are subjective, broad and significantly, can differ between patients and clinicians. Measures of performance status may fail to detect small, but meaningful changes in activity behaviours. Objective assessment of activity behaviours using accelerometers could provide a more reliable and sensitive method to assess physical activity and sedentary behaviour, particularly in advanced cancer populations. Objective assessment of activity behaviours using accelerometers has been demonstrated to accurately measure physical activity when compared to oxygen consumption. Triaxial accelerometry is considered the most accurate assessment for physical activity in chronic disease populations.

Preliminary research in patients with MPE indicates that patients have very low activity levels. Participants with MPE spent more that 70% of waking hours sedentary (i.e., activities of very low energy expenditure, sitting or lying down). Those patients with MPE with the best performance status and longest survival were significantly more active and less sedentary than those with a poor performance status and limited survival. However, these preliminary results require replication. Further, it is not yet known if activity behaviours are associated with quality of life or symptoms such as dyspnea in this patient population. Evidence from other cancer survivor populations suggests that activity behaviours are linked to quality of life and symptoms. In patients with breast, colorectal, lung and ovarian cancer, those that are more physically active report better quality of life. In patients with lung cancer, symptoms such as breathlessness and fatigue appear to be associated with lower physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an MPE (i.e. one in which malignant cells are identified in the pleural fluid or pleural biopsy); or a large exudative pleural effusion without other causes in a patient with known disseminated extra-thoracic malignancy

Exclusion Criteria:

* Patients with Age <18 years; pleural infection; pregnant or lactating; inability to consent or comply with the protocol; anticipated pleural drainage procedure within one week subsequent to recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an MPE
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Activity Behaviours (vertical axis movement counts per min) | 7 days
  Recorded objectively by a triaxial accelerometer (ActiGraph GT3X+ Pensacola, FL, USA).
Quality of life (in mm) | 7 days
  Assessed by a 100 mm visual analogue scale with "the best imaginable health state" at 0 mm and "the worst imaginable health state" at 100 mm
Respiratory symptoms (in mm) | 7 days
  Assessed by a 100 mm visual analogue scale with "no breathlessness" at 0 mm and "worst breathlessness imaginable" at 100 mm.
Survival (in number of days) | 12 months
  Recorded from date of Actigraph initialization to death or 12-month, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: David CL Lam, PhD, MD, Principal Investigator — University of Hong Kong Queen Mary Hospital
Locations (1):
- University of Hong Kong Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clive AO, Kahan BC, Hooper CE, Bhatnagar R, Morley AJ, Zahan-Evans N, Bintcliffe OJ, Boshuizen RC, Fysh ET, Tobin CL, Medford AR, Harvey JE, van den Heuvel MM, Lee YC, Maskell NA. Predicting survival in malignant pleural effusion: development and validation of the LENT prognostic score. Thorax. 2014 Dec;69(12):1098-104. doi: 10.1136/thoraxjnl-2014-205285. Epub 2014 Aug 6. PMID 25100651
- [Background] Thomas R, Francis R, Davies HE, Lee YC. Interventional therapies for malignant pleural effusions: the present and the future. Respirology. 2014 Aug;19(6):809-22. doi: 10.1111/resp.12328. Epub 2014 Jun 19. PMID 24947955
- [Background] Owen N. Sedentary behavior: understanding and influencing adults' prolonged sitting time. Prev Med. 2012 Dec;55(6):535-9. doi: 10.1016/j.ypmed.2012.08.024. Epub 2012 Sep 8. PMID 22968124
- [Background] Kelly LA, McMillan DG, Anderson A, Fippinger M, Fillerup G, Rider J. Validity of actigraphs uniaxial and triaxial accelerometers for assessment of physical activity in adults in laboratory conditions. BMC Med Phys. 2013 Nov 26;13(1):5. doi: 10.1186/1756-6649-13-5. PMID 24279826
- [Background] Van Remoortel H, Giavedoni S, Raste Y, Burtin C, Louvaris Z, Gimeno-Santos E, Langer D, Glendenning A, Hopkinson NS, Vogiatzis I, Peterson BT, Wilson F, Mann B, Rabinovich R, Puhan MA, Troosters T; PROactive consortium. Validity of activity monitors in health and chronic disease: a systematic review. Int J Behav Nutr Phys Act. 2012 Jul 9;9:84. doi: 10.1186/1479-5868-9-84. PMID 22776399
- [Background] Jeffery E, Lee YG, McVeigh J, Straker L, Wooding T, Newton RU, Peddle-McIntyre C. Feasibility of objectively measured physical activity and sedentary behavior in patients with malignant pleural effusion. Support Care Cancer. 2017 Oct;25(10):3133-3141. doi: 10.1007/s00520-017-3721-9. Epub 2017 Apr 28. PMID 28455548
- [Background] Vallance JK, Boyle T, Courneya KS, Lynch BM. Associations of objectively assessed physical activity and sedentary time with health-related quality of life among colon cancer survivors. Cancer. 2014 Sep 15;120(18):2919-26. doi: 10.1002/cncr.28779. Epub 2014 Jun 4. PMID 24898175
- [Background] Solberg Nes L, Liu H, Patten CA, Rausch SM, Sloan JA, Garces YI, Cheville AL, Yang P, Clark MM. Physical activity level and quality of life in long term lung cancer survivors. Lung Cancer. 2012 Sep;77(3):611-6. doi: 10.1016/j.lungcan.2012.05.096. Epub 2012 Jun 6. PMID 22681871
- [Background] Sloan JA, Cheville AL, Liu H, Novotny PJ, Wampfler JA, Garces YI, Clark MM, Yang P. Impact of self-reported physical activity and health promotion behaviors on lung cancer survivorship. Health Qual Life Outcomes. 2016 Apr 29;14:66. doi: 10.1186/s12955-016-0461-3. PMID 27129406
- [Background] Lynch BM, Cerin E, Owen N, Hawkes AL, Aitken JF. Prospective relationships of physical activity with quality of life among colorectal cancer survivors. J Clin Oncol. 2008 Sep 20;26(27):4480-7. doi: 10.1200/JCO.2007.15.7917. PMID 18802160
- [Background] Canario AC, Cabral PU, de Paiva LC, Florencio GL, Spyrides MH, Goncalves AK. Physical activity, fatigue and quality of life in breast cancer patients. Rev Assoc Med Bras (1992). 2016 Jan-Feb;62(1):38-44. doi: 10.1590/1806-9282.62.01.38. PMID 27008491
- [Background] Beesley VL, Price MA, Butow PN, Green AC, Olsen CM; Australian Ovarian Cancer Study Group; Australian Ovarian Cancer Study - Quality of Life Study Investigators; Webb PM. Physical activity in women with ovarian cancer and its association with decreased distress and improved quality of life. Psychooncology. 2011 Nov;20(11):1161-9. doi: 10.1002/pon.1834. Epub 2010 Aug 26. PMID 20740686
- [Background] Cheville AL, Novotny PJ, Sloan JA, Basford JR, Wampfler JA, Garces YI, Jatoi A, Yang P. The value of a symptom cluster of fatigue, dyspnea, and cough in predicting clinical outcomes in lung cancer survivors. J Pain Symptom Manage. 2011 Aug;42(2):213-21. doi: 10.1016/j.jpainsymman.2010.11.005. Epub 2011 Mar 12. PMID 21398089
- [Background] O'Driscoll M, Corner J, Bailey C. The experience of breathlessness in lung cancer. Eur J Cancer Care (Engl). 1999 Mar;8(1):37-43. doi: 10.1046/j.1365-2354.1999.00129.x. PMID 10362952
- [Background] Fysh ET, Thomas R, Read CA, Kwan BC, Yap E, Horwood FC, Lee P, Piccolo F, Shrestha R, Garske LA, Lam DC, Rosenstengel A, Bint M, Murray K, Smith NA, Lee YC. Protocol of the Australasian Malignant Pleural Effusion (AMPLE) trial: a multicentre randomised study comparing indwelling pleural catheter versus talc pleurodesis. BMJ Open. 2014 Nov 6;4(11):e006757. doi: 10.1136/bmjopen-2014-006757. PMID 25377015
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Light RW, Rogers JT, Cheng D, Rodriguez RM. Large pleural effusions occurring after coronary artery bypass grafting. Cardiovascular Surgery Associates, PC. Ann Intern Med. 1999 Jun 1;130(11):891-6. doi: 10.7326/0003-4819-130-11-199906010-00004. PMID 10375337